CLINICAL TRIAL: NCT02370433
Title: Use of Prokinetics During Inpatient Bowel Care for SCI Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dr. Mark Korsten, Chief of Gastroneterology, James J. Peters Veterans Affairs Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: KOR-12-035
Record Dates: First submitted 2015-02-18; First posted 2015-02-25 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Spinal Cord Injury; Neurogenic Bowel
Keywords: Spinal Cord Injury; Neurogenic Bowel; Bowel Evacuation
MeSH Terms: conditions — Spinal Cord Injuries; Neurogenic Bowel | interventions — Glycopyrrolate

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (3):
- Bowel Evacuation via IV (Experimental): The study design will consist of an intravenous (IV) screening visit to determine each individual's response to neostigmine and glycopyrrolate (NG).
  Interventions: Drug: Intravenous Neostigmine and Glycopyrrolate
- Bowel Evacuation Titration (Experimental): This design will consist of a dose titration for those subjects who respond positively to IV. These subjects will receive either a low dose and/or a high dose of NG via iontophoresis to determine their responsiveness.
  Interventions: Drug: Transdermal Neostigmine and Glycopyrrolate
- Bowel Evacuation Iontophoresis (Experimental): This design will consist of the incorporation of iontophoresis administration into clinical bowel care. The subject will receive the exact dose they responded to during the titration 3x per week for 2weeks.
  Interventions: Drug: Transdermal Neostigmine and Glycopyrrolate

INTERVENTIONS:
Drug: Intravenous Neostigmine and Glycopyrrolate
  Arms: Bowel Evacuation via IV
Drug: Transdermal Neostigmine and Glycopyrrolate
  Arms: Bowel Evacuation Iontophoresis; Bowel Evacuation Titration

SUMMARY:
Bowel care (BC) is a time-consuming and cumbersome activity of daily living for most individuals with SCI. Previous studies have reported that the average time to complete a BC routine is 45 minutes; 10-20% of SCI individuals report BC routines lasting for more than 1 hour. In past studies, the investigators have shown that a medication called neostigmine can increase bowel activity and thus, promote bowel movement. The investigators have successfully used this medication with traditional and novel methods of colonoscopic preparations, and have shown that it improves the quality of these preparations. In this study, we would like to test the applicability of this medication to bowel care routines.

The investigators believe that the addition of this medication to the beginning of regular bowel regiments will significantly decrease the time and effort needed to complete BC, thus improving patient perception of their BC routines and quality of life. SCI individuals followed by the James J Peters VA Medical Center (JJPVAMC) SCI Medical Service are admitted on a routine basis for inpatient respite care, therapy, and/or annual physicals. Such inpatient stays typically range in duration from 1 week to 3 weeks, during which the patient undergo BC routines assisted by the inpatient care team. BC routines are typically performed every other day, or thrice weekly (Monday, Wednesday, Friday) in "Blue Rooms" located on the inpatient SCI wards (IE and ID). The bowel care routine, including duration of procedure, use of assistive medications or devices, and completeness of bowel care are documented in the patients' electronic medical chart (CPRS) by care providers. The investigators propose to perform the described protocol in individuals who have been admitted to the hospital for routine care and are otherwise healthy. In doing so, the investigators can ensure that patients are vigilantly monitored during each BC session, and that any changes in BC pattern are accurately observed and documented. Furthermore, by performing these procedures on an inpatient basis, study investigators can ensure the consistency of care and daily routine, allowing for better control of study conditions.

DETAILED DESCRIPTION:
Part 1: IV Screening Twenty subjects with chronic SCI (>1 year) and difficulty with evacuation (DWE) managed by a regular, thrice weekly BC routines will be recruited for study participation. In order to determine eligibility for the study, the subject will have to undergo an IV screening to test whether or not they are responsive to the drug treatment (neostigmine-glycopyrrolate). If the subject responds (bowel movement) to the IV treatment, they will be allowed to continue on to part 2 of the study. If patient does not have a successful bowel movement, then they will be considered a non-responder and study participation will be discontinued.

Part 2: Baseline and Dose Titration Once eligibility has been determined, and subject consent has been obtained, each subject will undergo 1 week of baseline observation after admission. An abdominal x-ray (KUB) will be performed, the SCI Bowel Survey and Treatment Satisfaction Questionnaire (TSQM) will be administered, and the subject's weight determined. Each subject will continue with regular bowel care as an inpatient, and after 1 week, all of the baseline measurements (KUB, weight and surveys) will be repeated. This will be followed by a 2 visit- dose titration study of concomitantly administered, transcutaneous neostigmine methylsulfate (NEO) and glycopyrrolate (GLY). Each visit will be scheduled on a BC day. All procedures will take place in the "Blue Room" located in the SCI inpatient ward. Subjects will be prone throughout the duration of the study, in a stretcher routinely used during bowel care. As part of the setup, subjects will be instrumented with blood pressure cuff; intravenous access will be obtained at a peripheral vein (if one is not available), as a precautionary measure, since the drug will be administered via an Iontophoresis transdermal patch. Heart rate will be continuously monitored throughout the procedure through finger oximetry. Symptoms will be assessed every 5 minutes for the first 30 minutes, and then at 1 hour post drug administration. Once the subject has a positive response to one of the two doses, or the higher dose has been performed, the dose titration will be stopped. If the subject has a positive response (bowel movement within 60 minutes of drug administration) he/she will be eligible to continue to the third study phase. If the subject does not respond to either dose, the subject will be considered a non-responder and study participation will be discontinued. We expect that about 1/3rd of the subjects will be non-responders, or will be lost to attrition; therefore, we are prepared to over-recruit by 5 subjects in order to ensure that at least 15 subjects will be eligible to complete the second part of the study.

The study will be stopped once the patient experiences a bowel movement within 30 minutes of administering ION NEO because the protocol objective will have been achieved. If the patient should experience cardiopulmonary side effects when receiving the ION NEO on the lower doses that are not effectively reversed by the ION GLY, the study will be stopped. In addition, the study investigators reserve the right to stop the study should they have any other safety concerns.

Part 3: 2 Week Treatment Each subject will be assessed for their perception of their current BC routine using the Treatment Satisfaction Questionnaire for Medication (TSQM-Appendix 1), and their bowel habits using the bowel survey (Appendix 2).The subject will then be asked to continue with their normal BC routine for two weeks during their inpatient stay, with the exception that NEO and GLY will be administered at the beginning of each BC session as an adjunct to each subject's normal routine. Each BC session will be documented by a study team member including the time needed to complete BC, methods used (i.e. number of enemas used, oral laxatives, suppositories, digital stimulation, abdominal massage) and the quality and completeness of the bowel movement. Heart rate, oxygenation and blood pressure will be monitored continuously. Subjects will be weighed at baseline, once after each week of treatment and once at the post treatment follow-up visit. After two weeks of treatment, each subject will undergo a final KUB and be reassessed for their perception of the BC routine for the past two weeks using the TSQM and their bowel habits (bowel survey).

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-75 years
* Spinal Cord Injury (SCI):
* greater than 1 year duration
* excess time for bowel evacuation (> 60minutes per session)

Exclusion Criteria:

* Previous Adverse Reaction or Hypersensitivity to Electrical Stimulation
* Do not require additional bowel care or have "normal bowel function"
* Known sensitivity to Neostigmine and Glycopyrrolate
* Blockage in Bowel and/or Bladder
* Myocardial Infarction in the past 6months
* Blood Pressure ≥160/100 mmHg with/without being on 3 or more different classes of antihypertensive medications
* Organ Damage (heart & kidney) and/or transient ischemic attack (TIA)- cerebrovascular accident (CVA) as a result of hypertension
* Known past history of coronary artery disease, chronic heart failure, bradyarrythmia
* Slow Heart Rate (<45bpm)
* Active respiratory diseases
* Known history of asthma during lifetime
* Recent (within 3months) respiratory infections
* Adrenal Insufficiency
* Pregnancy or potential for pregnancy
* Lactating/nursing females
* Use of any antibiotics in past 7days
* Use of medications known to affect respiratory system
* Concurrent participation in other clinical trials (within 30days)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-12; Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Biological Response to Study Medication (Changes in BC habits (time to complete BC, reductions/ increases in secondary methods (enemas, suppositories, oral supplements) needed to complete BC will be assessed) | 24months
  We aim to evaluate the effect of treatment with NG through Iontophoresis during routine bowel care (BC) during inpatient visits. Changes in BC habits (time to complete BC, reductions/ increases in secondary methods (enemas, suppositories, oral supplements) needed to complete BC will be assessed

SECONDARY OUTCOMES:
Effect of Medication on Impaction (changes in fecal impaction and constipation by documenting weekly weight and pre to post treatment plain abdominal x-ray) | 24months
  We aim to To evaluate changes in fecal impaction and constipation by documenting weekly weight and pre to post treatment plain abdominal x-ray
Subjective Feedback from Inpatients (Treatment Satisfaction Questionnaire for Medication (TSQM) | 24months
  We aim To compare patient perception of the proposed treatment using the Treatment Satisfaction Questionnaire for Medication (TSQM) before and after the inpatient treatment period.

CONTACTS AND LOCATIONS:
Locations (1):
- James J. Peters VA Medical Center, The Bronx, New York, United States